CLINICAL TRIAL: NCT00499720
Title: Expanded Access Program for Aztreonam Lysine for Inhalation in Patients With Cystic Fibrosis and Pseudomonas Aeruginosa Airway Infection Who Have Limited Treatment Options and Are at Risk for Disease Progression
Brief Title: Aztreonam Lysine for Inhalation in Patients With Cystic Fibrosis and Pseudomonas Aeruginosa Airway Infection
Status: Approved for marketing | Type: Expanded Access
Sponsor: Gilead Sciences (Industry)
Responsible Party: Debra Cibene/Senior Clinical Research Associate, Gilead Sciences, Inc.
Other Study IDs: EA-US-205-0111
Record Dates: First submitted 2007-07-09; First posted 2007-07-11 (Estimated); Last update posted 2011-08-02 (Estimated); Status verified 2011-07

CONDITIONS: Cystic Fibrosis; Pseudomonas Aeruginosa Airway Infection
Keywords: Cystic Fibrosis; Pseudomonas aeruginosa; airway infection; Aztreonam Lysine for Inhalation
MeSH Terms: conditions — Cystic Fibrosis; Pseudomonas Infections | interventions — Inhalation

INTERVENTIONS:
Drug: Aztreonam Lysine for Inhalation — 75 mg three times a day via inhalation for 28 days followed by 28 days off drug.

SUMMARY:
The primary objective of this program is to provide expanded access to aztreonam lysine for inhalation (AZLI) 75 mg prior to its commercial availability to patients with cystic fibrosis (CF) and chronic P. aeruginosa airway infection who have limited treatment options and are at risk for disease progression.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be eligible for participation in this study:

* ≥ 6 years of age
* Subject has CF as diagnosed by one of the following:

  * Documented sweat chloride ≥ 60 mEq/L by quantitative pilocarpine iontophoresis test
  * Two well characterized genetic mutations in the CFTR gene
  * Abnormal nasal potential difference with accompanying symptoms characteristic of CF
* At high risk for disease progression as defined by one of the following subject populations:

  * First Cohort Criteria:

    * Those who are wait listed or eligible for lung transplant based on FEV1 criteria. Patients who have a level of lung function impairment consistent with lung transplantation criteria, but who are ineligible for transplantation for other reasons, can enroll in this program; or
    * Completed participation in CP-AI-006 (through Visit 20). Subjects who withdraw from CP-AI-006 prior to completing all courses of AZLI and all study visits will not be eligible for this protocol.
  * Second Cohort Criteria:

    * Meets first cohort criteria
    * FEV1 ≤ 40% predicted at the time of consent
  * Third Cohort Criteria:

    * Meets first or second cohort criteria
    * FEV1 ≤ 50% predicted at the time of consent

Exclusion Criteria:

Subjects who meet any of the following exclusion criteria are not to be enrolled in this study:

* Subjects with any serious or active medical or psychiatric illness that, in the opinion of the investigator, would interfere with subject treatment, assessment or compliance with the protocol or dosing requirements
* Subjects with hypersensitivity to any of the components of the drug product
* Currently enrolled in another clinical trial
* Pregnant or lactating females

Min Age: 6 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (57):
- United States (56):
  - Birmingham, Alabama
  - Anchorage, Alaska
  - Phoenix, Arizona
  - Little Rock, Arkansas
  - Los Angeles, California
  - Sacramento, California
  - San Francisco, California
  - Denver, Colorado
  - Hartford, Connecticut
  - Ft, Meyers, Florida
  - Gainesville, Florida
  - Orlando, Florida
  - St. Petersburg, Florida
  - Tampa, Florida
  - Boise, Idaho
  - Chicago, Illinois
  - Maywood, Illinois
  - Des Moines, Iowa
  - Wichita, Kansas
  - New Orleans, Louisiana
  - Boston, Massachusetts
  - Detroit, Michigan
  - Minneapolis, Minnesota
  - Columbia, Missouri
  - Kansas City, Missouri
  - Great Falls, Montana
  - Las Vegas, Nevada
  - Long Branch, New Jersey
  - New Brunswick, New Jersey
  - Albuquerque, New Mexico
  - Albany, New York
  - Buffalo, New York
  - New Hyde Park, New York
  - New York, New York
  - Syracuse, New York
  - Valhalla, New York
  - Chapel Hill, North Carolina
  - Akron, Ohio
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Toledo, Ohio
  - Oklahoma City, Oklahoma
  - Hershey, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Sioux Falls, South Dakota
  - Memphis, Tennessee
  - Dallas, Texas
  - Fort Worth, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Norfolk, Virginia
  - Portsmouth, Virginia
  - Richmond, Virginia
  - Seattle, Washington
- San Juan, Puerto Rico